CLINICAL TRIAL: NCT06907602
Title: Optimizing Neoadjuvant Treatment Regimens for Locally Advanced Esophageal Squamous Cell Carcinoma: A Phase II Clinical Study
Brief Title: Optimizing Neoadjuvant Treatment Regimens for Locally Advanced Esophageal Squamous Cell Carcinoma
Acronym: ONTRESCC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Military 301 Hospital (Unknown); Peking University Cancer Hospital & Institute (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Keypoint 002
Record Dates: First submitted 2025-03-27; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; neoadjuvant chemoimmunotherapy; radiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Drug Therapy; Immunotherapy; pembrolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 2 cycles chemoimmunotherapy plus surgery (Experimental): 2 cycles chemoimmunotherapy and surgery
  Interventions: Drug: Chemotherapy; Drug: Immunotherapy (Pembrolizumab)
- 4 cycles chemoimmunotherapy plus surgery (Experimental): 4 cycles chemoimmunotherapy and surgery
  Interventions: Drug: Chemotherapy; Drug: Immunotherapy (Pembrolizumab)
- 4 cycles chemoimmunotherapy plus radiotherapy and surgery (Experimental): 4 cycles chemoimmunotherapy plus radiotherapy and surgery
  Interventions: Drug: Chemotherapy; Drug: Immunotherapy (Pembrolizumab); Radiation: radiotherapy

INTERVENTIONS:
Drug: Chemotherapy — carboplatin plus nab-paclitaxel
Drug: Immunotherapy (Pembrolizumab) — Pembrolizumab
Radiation: radiotherapy — 40-45Gy/20fx，5 times a week
  Arms: 4 cycles chemoimmunotherapy plus radiotherapy and surgery

SUMMARY:
Our previous study, a single-center, prospective, single-arm Phase II study (Keypoint001) has demonstrated the efficacy and safety of neoadjuvant chemotherapy combined with immunotherapy in locally advanced (cT3-4N+M0) esophageal squamous cell carcinoma. The results show that the pathological complete response rate (pCR) reaches 35%, and the major pathological response rate is over 70%, which is much higher than that of patients receiving chemotherapy alone. Meanwhile, no severe adverse drug reactions have been found in terms of safety, so this treatment regimen is safe and reliable.

However, the cycle of neoadjuvant immunotherapy is still under exploration. Currently, the mainstream research centers adopt a regimen of 2 to 4 cycles. The exploration results of our center have found that most patients' conditions can be further alleviated after 4 cycles compared with after 2 cycles, but there are still a small number of patients with no obvious remission. Therefore, we consider observing whether patients with no obvious remission can achieve a better pathological response rate through further radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* Age ≥ 18 years old
* Pathological confirmation of esophageal squamous cell carcinoma
* Endoscopic ultrasound, enhanced CT scan of the neck, chest, and abdomen, and esophageal magnetic resonance imaging evaluate as T3 or resectable T4 PET/CT、 Cervical, thoracic, and abdominal enhanced CT evaluation of N0 or N+
* No clear distant metastasis (M0) and only cervical or supraclavicular lymph node metastasis (M1a)
* Tumor longitudinal diameter ≤ 10cm
* The tumor did not involve the dentate line
* ECOG score 0 or 1
* No hematological diseases, no liver or kidney dysfunction
* Absolute neutrophil count ≥ 1.5 × 109/L
* Platelets ≥ 100 × 109/L
* Hemoglobin ≥ 11g/L
* ALT ≤ 2 times the upper limit of normal value
* TBil ≤ 1.5 times the upper limit of normal value
* Creatinine clearance rate (Cockroft) ≥ 50ml/min
* Obtain informed consent

Exclusion Criteria:

* T staging evaluation is T1/T2
* PET/CT and other evaluations show distant metastasis (M1)
* Planned pregnancy or patients during pregnancy or lactation
* History of previous chemotherapy, radiation therapy, or immunotherapy
* Previous severe coronary heart disease and heart failure (NYHA grade III/IV)
* Previous pulmonary interstitial fibrosis or severe pulmonary dysfunction that cannot tolerate surgery
* Previous autoimmune disease requiring systemic treatment within 2 years
* Previous immunodeficiency diseases or the need for systemic steroid replacement therapy
* Previous motor or sensory neurotoxic diseases
* Previous mental illness
* Potential diseases that may affect patients' ability to receive planned treatment, such as drug allergies
* Acute infectious diseases requiring systemic treatment
* Previous HIV, HBV, or HCV infections
* Previously received stem cell or solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological response | After surgery
  Postoperative pathology according to CAP classification.
2-year and 5-year overall survival | 2 years and 5 years after therapy
  overall survival after 2 years and 5 years

SECONDARY OUTCOMES:
Adverse effect incidence | 1 years after therapy
  Adverse effect according to CTCAE and RTOG criteria
R0 resection rate | After surgery
postoperative complications | After surgery
  postoperative complications according to Clavien-Dindo classification
2-year and 5-year disease-free survival | 2 years and 5 years after therapy
  disease-free survival after 2 years and 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided